CLINICAL TRIAL: NCT06257420
Title: Low Dose Rapamycin in ME/CFS, Long-COVID, and Other Infection Associated Chronic Conditions
Status: Enrolling by invitation | Type: Observational
Sponsor: Simmaron Research Inc. (Other)
Collaborators: Center For Complex Diseases-Seattle, WA (Unknown); Sierra Internal Medicine, Incline Village, NV (Unknown); Center for Complex Diseases- Palo Alto, CA (Unknown); Simmaron Research Inc. R&D Lab, University of Wisconsin, Milwaukee (UWM) (Unknown); Bateman Horne Center, Salt Lake City, UT (Unknown); Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: SRI-RP-2023-1
Record Dates: First submitted 2024-01-17; First posted 2024-02-14 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Myalgic Encephalomyelitis; Long-COVID
Keywords: ME/CFS; Long-COVID; Infection Associated Chronic Conditions
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Post-Acute COVID-19 Syndrome | interventions — Sirolimus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood will be collected to isolate plasma, PBMC, serum and RNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ME/CFS and Long-COVID patients with serological evidence of autophagy disruption: ME/CFS and Long-COVID patients with serological evidence of autophagy disruption at baseline will be prescribed once weekly rapamycin at a max dose of 6mg per week.
  Interventions: Drug: Rapamycin
- ME/CFS and Long-COVID patients without serological evidence of autophagy disruption: ME/CFS and Long-COVID patients without serological evidence of autophagy disruption at baseline will be prescribed once weekly rapamycin at a max dose of 6mg per week.
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin — Once weekly oral rapamycin
  Other Names: Sirolimus; Rapamune

SUMMARY:
The goal of this observational study is to assess the clinical response and the effect of autophagy function in patients before, during and throughout oral low dose sirolimus (rapamycin) therapy. The main questions this study aims to answer are:

* Does rapamycin reduce the overall symptom burden in this patient population and does it improve the quality of life?
* Does rapamycin change mTOR driven autophagy deficits observed in a subset of patients?

Participants will be asked to complete a series of questionnaires and quality of life instruments before starting rapamycin therapy prescribed by their physician and throughout their course of treatment. Study blood samples will be collected before starting therapy and throughout the course of treatment to assess serological markers of autophagy function.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ME/CFS that meets the Institute of Medicine (IOM) criteria
* Diagnosis of Long-COVID (PASC clinical criteria)

Exclusion Criteria:

* No diagnosis of ME/CFS or Long-COVID

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are recruited by study clinicians who are Principal Investigators in this trial.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2025-12-11 (Estimated); Study Completion 2026-06-11 (Estimated)

PRIMARY OUTCOMES:
The Short Form (36) Health Survey | 1 year
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Multidemensional Fatigue Inventory (MFI) | 1 year
  The MFI is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue.
The Bell Activity Scale | 1 year
  The Bell CFIDS Disability Scale is described in the book, The Doctor's Guide to Chronic Fatigue Syndrome: Understanding, Treating and Living with CFIDS (Bell 1995). This scale assesses functional ability in adult ME/CFS patients. Eleven statements describe patient status such as level of symptoms at rest, level of symptoms with exercise, activity level, and ability to perform work, travel and self care.

SECONDARY OUTCOMES:
Change in mTOR activation panel and blood markers involved in autophagy function. | 1.5 year
  Change in concentrations of phosphorylated autophagy-related gene proteins in blood

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Gottschalk, PhD, Principal Investigator — Simmaron Research Inc.
Locations (5):
- United States (5):
  - Center For Complex Diseases, Palo Alto, California
  - The Mayo Clinic, Rochester, Minnesota
  - Sierra Internal Medicine, Incline Village, Nevada
  - Bateman Horne Center, Salt Lake City, Utah
  - Center For Complex Diseases, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
IPD will be available to share with non-profit and academic institutions.

REFERENCES:
- [Background] Gottschalk G, Peterson D, Knox K, Maynard M, Whelan RJ, Roy A. Elevated ATG13 in serum of patients with ME/CFS stimulates oxidative stress response in microglial cells via activation of receptor for advanced glycation end products (RAGE). Mol Cell Neurosci. 2022 May;120:103731. doi: 10.1016/j.mcn.2022.103731. Epub 2022 Apr 26. PMID 35487443
- [Background] Gottschalk CG, Whelan R, Peterson D, Roy A. Detection of Elevated Level of Tetrahydrobiopterin in Serum Samples of ME/CFS Patients with Orthostatic Intolerance: A Pilot Study. Int J Mol Sci. 2023 May 13;24(10):8713. doi: 10.3390/ijms24108713. PMID 37240059
- See also: Simmaron Website — http://www.simmaron.com